CLINICAL TRIAL: NCT04067310
Title: Randomized, Open-label Study Using Spray Skin Protector Versus Conventional Treatment to Prevent Acute Radiodermatitis in Patients With Anal and Rectal Canal Cancer.
Brief Title: Study Using Spray Skin Protector Versus Conventional Treatment to Prevent Acute Radiodermatitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Fabiana Verdan Simões, Principal Research Nurse, Instituto Nacional de Cancer, Brazil
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PROT
Record Dates: First submitted 2019-08-20; First posted 2019-08-26 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Radiodermatitis; Injury, Radiation
Keywords: barrier film; spray skin protection; liquid-film; barrier product
MeSH Terms: conditions — Radiodermatitis; Radiation Injuries

STUDY DESIGN:
Intervention Model Description: After signing the Informed Consent Form, randomization will be carried out in two groups: Experimental, which will use the skin protector in spray and control, which will use the moisturizer Dnativ Revita Derm.
Who Masked: Outcomes Assessor
Masking Description: Blinding will be in skin evaluation and statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Experimental (Experimental): Participants who will use the spray skin protector
  Interventions: Other: Spray skin protector
- Group control (Active Comparator): Participants who will use moisturizer Dnativ Revita Derm.
  Interventions: Other: moisturizer Dnativ Revita derm

INTERVENTIONS:
Other: Spray skin protector — Patients will use spray skin protector treatment from the randomization day until the last day of radiotherapy.
  Other Names: barrier film to prevent radiodermatitis
  Arms: Group Experimental
Other: moisturizer Dnativ Revita derm — Patients will use conventional preventive treatment from the randomization day until the last day of radiotherapy.
  Other Names: conventional treatment to prevent radiodermatitis
  Arms: Group control

SUMMARY:
This is a randomized, open-label, single-institution trial designed to evaluate the effectiveness of a spray skin protector in preventing moist desquamation caused by radiotherapy treatment.

This technology, spray skin protection, depending on the manufacturer, is primarily intended to prevent or reduce contact dermatitis. However, this study will be evaluated for use in preventing moist desquamation caused by ionizing radiation. The comparing agent will be a moisturizer, agreed upon at the local Institution of the study for use in the prevention of radiodermatitis. As secondary objectives: describe adverse events, diarrhea, pain and pruritus.

The study will be conducted at the radiotherapy outpatient clinic of the Cancer Hospital I (HCI) of National Cancer Institute (INCA) in Brazil.

DETAILED DESCRIPTION:
The hypotheses are:

Null (Ho): The incidence of moist desquamation with the spray skin protector is greater than or equal to the incidence of moist desquamation in the control group.

Alternative (H1): The incidence of moist desquamation with the spray skin protector is lower than the incidence of moist desquamation in the control group.

The evaluation of the skin of the participants will be weekly, with blinding of this professional. For the evaluation of secondary objectives, adverse events will be applied in the assessment scales of diarrhea, pruritus and pain by the CTCAE version 5.0; and the burning or burning sensation will be recorded only.

ELIGIBILITY:
Inclusion Criteria: patients with anal and rectal cancer with indication for radiotherapy and conventional fractionation of treatment in a linear accelerator; age > or = 18 years; no previous history of radiotherapy in the same field/site of treatment (reirradiation).

-

Exclusion Criteria:patients with pre-existing irradiated dermatitis, which makes skin assessment difficult; previous report of allergic reaction to any of the products used in the research.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabiana V Simões, Principal Investigator — Universidade Federal do Rio de Janeiro (UFRJ); Rafael C Silva, Principal Investigator — Universidade Federal do Rio de Janeiro (UFRJ); Beatriz G R B Oliveira, Principal Investigator — Universidade Federal Fluminense (UFF)
Locations (1):
- INCA Research Center, Rio de Janeiro, Rio de Janeiro, Brazil

RESULTS

PARTICIPANT FLOW:
Groups:
- Group Experimental: Participants who used the skin protector spray
  Skin protector spray: Patients used skin protector spray treatment from the randomization day until the last day of radiotherapy.
- Group Control: Participants who will use moisturizer Dnativ Revita Derm.
  Moisturizer Dnativ Revita derm: Patients used conventional preventive treatment from the randomization day until the last day of radiotherapy.
Period: Overall Study
Arm/Group | Group Experimental | Group Control
Started | 36 | 36
Completed | 31 | 29
Not Completed | 5 | 7
Not completed — Physician Decision | 2 | 6
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group Experimental; Group Control: Intention to treat
- Total: Total of all reporting groups
Arm/Group | Group Experimental | Group Control | Total
Number analyzed (Participants) | 34 | 29 | 63
Age, Customized [Count of Participants; unit: Participants]
  21-66 | 19 | 17 | 36
  67-90 | 15 | 12 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 15 | 9 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 14 | 23
  Black | 3 | 6 | 9
  Brown | 22 | 8 | 30
  Indigenous | 0 | 1 | 1
  Asian | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 34 | 29 | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Categorized by RTOG Grading Scale
Description: RTOG ACUTE Radiation Morbidity - Tissue: Skin
  * Grade 1: Follicular, faint or dull erythema / epilation / dry desquamation / decreased sweating;
  * Grade 2: Tender or bright erythema, patchy moist desquamation / moderate edema;
  * Grade 3: Confluent, moist desquamation other than skin folds, pitting edema;
  * Grade 4: Ulceration, hemorrhage, necrosis.
Time Frame: From the first day of radiotherapy up to eight weeks
Population: Patients with anal canal or rectum cancer with indication for RT and conventional treatment fractionation in Linear Accelerator (< 250cGy/day); 18+ years old; no previous history of radiotherapy in the same treatment field/site (reirradiation); with no preexisting dermatitis at the irradiated site that would make it difficult to assess the skin; and no previous report of allergic reaction to any products used in the research.
Measure: Count of Participants; unit: Participants
Groups:
- Group Experimental: Maximum RTOG grade - Intention to Treat:
  Grade 1 - 12 (35.3%) Grade 2 - 11 (32.4%) Grade 3 - 10 (29.4%) Grade 4 - 1 (2.9%)
- Group Control: Maximum RTOG grade - Intention to Treat:
  Grade 1 - 6 (20.7%) Grade 2 - 11 (37.9%) Grade 3 - 11 (37.9%) Grade 4 - 1 (3.4%)
Arm/Group | Group Experimental | Group Control
Number analyzed (Participants) | 34 | 29
Participants
  RTOG Grade 1 | 12 | 6
  RTOG Grade 2 | 11 | 11
  RTOG Grade 3 | 10 | 11
  RTOG Grade 4 | 1 | 1

2. Secondary Outcome: Adverse Events
Description: Occurrence of adverse events after the beginning of radiotherapy
Time Frame: From the first day of radiotherapy up to eight weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group Experimental | Group Control
Number analyzed (Participants) | 34 | 29
Participants
  Body fluid losses before radiotherapy | 29 | 23
  Body fluid losses during radiotherapy | 33 | 28
  Relief | 14 | 12
  Discomfot | 5 | 2
  Stinging | 5 | 5
  Diarrhea | 7 | 12
  Fecal incontinence | 12 | 10
  Urinary incontinence | 16 | 11
  Fistula | 1 | 1
  Constipation | 1 | 5
  Herpes simplex | 1 | 1
  Adult Acute Respiratory Syndrome | 0 | 1
  Nausea | 2 | 2
  Urinary tract pain | 1 | 2

ADVERSE EVENTS:
Time Frame: From the first day of radiotherapy up to eight weeks
Arm/Group | Group Experimental | Group Control
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/34 | 1/29
Other Adverse Events (participants affected / at risk) | 33/34 | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group Experimental (N=34) | Group Control (N=29)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) — Severe Acute Respiratory Syndrome caused by SRAS-CoV-2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group Experimental (N=34) | Group Control (N=29)
Discomfort (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4)
Stinging (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5)
Body fluid losses before radiotherapy (Skin and subcutaneous tissue disorders) | 29 (29) | 23 (23)
Anal fistula (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Body fluid losses during radiotherapy (Skin and subcutaneous tissue disorders) | 33 (33) | 28 (28)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 12 (12)
Fecal incontinence (Gastrointestinal disorders) | 12 (12) | 10 (10)
Urinary incontinence (Renal and urinary disorders) | 16 (16) | 11 (11)
Constipation (Gastrointestinal disorders) | 1 (1) | 5 (5)
Herpes simplex reactivation (Infections and infestations) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
The small sample size was a methodological limitation. When the COVID-19 pandemic emerged, the institution reduced the number of vacancies in the regulation system for the radiotherapy outpatient clinic of the HCI-INCA. Other factor that hindered attracting participants was the opening of new vacancies for radiotherapy in other institutions that had been closed until then.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT04067310/Prot_SAP_000.pdf